CLINICAL TRIAL: NCT05750576
Title: Impact of ECMO Cannula Chlorhexidine-impregnated Dressings to Decrease Extracorporeal Membrane Oxygenation-cannula Related Infection Rate
Acronym: DRESSING-ECMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP190190; 2020-A02557-32 (Other: ID-RCB)
Record Dates: First submitted 2023-01-19; First posted 2023-03-01 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Cardiogenic Shock; Extracorporeal Membrane Oxygenation Complication; Acute Respiratory Distress Syndrome; Infections
Keywords: ECMO; Cardiogenic Shock; ARDS; Infection
MeSH Terms: conditions — Shock, Cardiogenic; Respiratory Distress Syndrome; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chlorhexidine-impregnated dressings (Experimental)
  Interventions: Device: Chlorhexidine-impregnated dressings
- Non impregnated dressings (Placebo Comparator)
  Interventions: Device: Non impregnated dressings

INTERVENTIONS:
Device: Chlorhexidine-impregnated dressings — Sterile adhesive transparent dressings impregnated with Chlorhexidine Gluconate gel applied to ECMO cannulae for up to 7 consecutive days for each dressing, in the absence of exudation or bleeding at the point of insertion and until explantation of the ECMO, sometimes requiring dressing changes.
  Arms: Chlorhexidine-impregnated dressings
Device: Non impregnated dressings — Single transparent adhesive dressings not impregnated with Chlorhexidine Gluconate applied to ECMO cannulae for up to 7 consecutive days for each dressing, in the absence of exudation or bleeding at the point of insertion and until explantation of the ECMO, sometimes requiring dressing changes.
  Arms: Non impregnated dressings

SUMMARY:
The Dressing-ECMO trial is a prospective, open-label, multicenter, controlled trial randomizing patients who received percutaneous ECMO to cannula chlorhexidine-impregnated dressing vs standard dressing. The study goal is to determine if cannula chlorhexidine-impregnated dressings can reduce the number of cannula major-related infections with or without bloodstream infection

DETAILED DESCRIPTION:
Open-label, multicenter, randomized, controlled trial. This study will be conducted in patients with cardiogenic shock or acute respiratory distress syndrome receiving percutaneous ECMO for less than 24h. All consecutive eligible patients will be proposed to participate. They will be randomly allocated in a 1:1 ratio to conventional cannula dressing, or cannula chlorhexidine-impregnated dressing, using an online, central randomisation service, to ensure allocation concealment. Blocked randomization will be performed using random block size. Randomization will be stratified according to center and ECMO type (i.e veno venous or arteriovenous). In both groups, peripheral blood sample will be cultured daily from first day on ECMO to 48h after ECMO removal, death on ECO or ECMO day 30 whichever occurs first. In case of ECMO cannula infection suspicion, deep samples of the cannula will be cultured according to the usual procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cardiogenic shock or refractory acute respiratory distress syndrome ECMO VA or VV ECMO for less than 24 hours.
* ECMO duration > 48 hours
* Obtained written informed consent from the trusted person or family member/relative. Depending on the emergency consent, randomization may take place and consent of the trusted person/relative/family will be obtained as soon as possible. The patient will be asked to give his/her consent for the continuation of the trial when hid/her condition will allow.
* Affiliation to a social security system (excluding state medical aid)

Exclusion Criteria:

* Age <18 years
* Initiation of ECMO for more than 24 hours
* Surgical (i.e. non percutaneous) cannulation
* Patient moribund on day of randomization, SAPS II >90
* Known allergy to chlorhexidine
* Antibiotic prophylaxis at ECMO cannulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence per 1000 ECMO days of ECMO cannula-related infection episodes, associated or not with bacteremia/fungemia | From ECMO initiation date (baseline) and up to day 60

SECONDARY OUTCOMES:
Colonization of ECMO cannulas at Day 7 and weaning from ECMO | Day 7 to 2 days after ECMO weaning date
Number of dressing changes for soiling or detachment | From day 1 to 2 days after ECMO weaning date
Number of days alive without antibiotics/fungal agents on ECMO | Between day 1 and Day 60
Total duration of ECMO | Between ECMO initiation date (baseline) and ECMO weaning date
Number of day in ICU | Between day 1 and Day 60
Overall survival | Day7, Day 30, Day 60
Cumulative incidence of ECMO cannula-related bacteremia/fungemia | From ECMO initiation date (baseline) and up to day 60
Cumulative incidence of each cannula infection endpoint in both arms | From ECMO initiation date (baseline) and up to day 60
Incidence of contact dermatitis or skin allergy | From ECMO initiation date (baseline) and up to day 60

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - CH Sud Francilien, Corbeil-Essonnes
  - Hôpital Henri-Mondor, Créteil
  - CHRU Nancy - Hôpitaux de Brabois, Nancy
  - Hôpital Pitié Salpêtrière, Paris
  - Hôpital Foch, Suresnes